CLINICAL TRIAL: NCT05278065
Title: Complimentary Electronic Cigarettes for Harm Reduction Among Adult Smokers With Asthma
Brief Title: E-cigarettes for Harm Reduction in Adults With Asthma
Acronym: SWAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Alexander Sokolovsky, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1908002509; P20GM130414 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-03-14 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Smoking; Asthma; Electronic Cigarette Use; Cigarette Smoking
Keywords: Smoking; Vaping; Cigarettes; E-cigarettes; electronic nicotine delivery systems; ENDS; Asthma; Substitution; pulmonary function; harm reduction
MeSH Terms: conditions — Smoking; Asthma; Vaping; Cigarette Smoking; Harm Reduction | interventions — Nicotine; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: 2:1 allocation of experimental to assessment only control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic cigarette (Experimental): Participants in this experimental condition will be provided with a 4th generation electronic cigarette device and disposable cartridges.
  Interventions: Other: Nicotine
- Smoking As Usual (No Intervention): Participants in this assessment-only condition will continue smoking as usual.

INTERVENTIONS:
Other: Nicotine — Participants will be provided with electronic cigarettes and 5% nicotine e-liquid cartridges for 8 weeks and encouraged at weekly assessments to use the electronic cigarette any time they would normally smoke. Participants will be able to choose commercially available e-liquid flavors (tobacco) at each weekly assessment.
  Other Names: electronic cigarette
  Arms: Electronic cigarette

SUMMARY:
Smoking is the main cause of preventable disease and death in the US and impacts respiratory illnesses including COPD and asthma. However, little is known about the effects on smoking and lung health of substituting cigarettes with ENDS in adults with asthma. This project aims to test whether providing ENDS to adults with asthma will lead to substitution of smoking for ENDS, reduced dependence, and improved lung function so such knowledge can inform interventions to reduce the public health burden of tobacco.

DETAILED DESCRIPTION:
This study will use an unequally allocated between-subjects (N=30) randomized, controlled design to investigate the influence of complimentary electronic nicotine delivery system (ENDS) provision on combustible cigarette and ENDS use, cigarette dependence, pulmonary function, clinical indicators and biomarkers, and substitution of smoking for ENDS use over 16 weeks. Participants will be adults from the local community with persistent asthma symptoms who are regular combustible cigarette smokers and do not also regularly use ENDS. The study will recruit 30 non-treatment seeking participants using flyers, advertisements, a website triaging visitors to the Center for Alcohol and Addiction Studies, and through targeted recruitment at community immunology clinic partners at Rhode Island Hospital as facilitated by mentor McQuaid. Participants meeting eligibility criteria will be assessed at baseline and then randomized to one of two study conditions: a complimentary ENDS provision condition or assessment-only control. Participants will return for eight weekly visits to complete follow-up assessments; participants in the experimental condition will be provided with additional e-liquid cartridges for their ENDS devices at all follow-up visits. Tobacco use behaviors (cigarette and ENDS) and lung function will be assessed at each visits, with additional collection of biological samples and assessments of nicotine dependence, self-efficacy for cessation, and mood at week eight. Provision of complimentary ENDS will discontinue eight weeks after enrollment. Participants will complete a remote follow-up assessment sixteen weeks after enrollment. This project, and all projects at the Center for Addiction and Disease Risk Exacerbation (CADRE) are supported by the Clinical Laboratory Core (CLC) which will oversee the collection and storage of data and biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (50%), 21 to 65 (inclusive) years of age;
* Persistent asthma symptoms (i.e., episodic symptoms of airflow obstruction / airway hyperresponsiveness (AHR) as documented in review of medical history);
* Currently prescribed SABA medication;
* Past-year smoking of ≥5 cigarettes/day;
* Exhaled CO ≥ 6 ppm at baseline;
* Zero breath alcohol during informed consent for participation;
* English-speaking at an 8th grade level.

Exclusion Criteria:

* Intention to quit smoking during the next 30 days;
* Current engagement in any smoking cessation treatment;
* Current self-identification as regular ENDS user or using ENDS > 2 days / week;
* Medical contraindication to nicotine;
* Pregnancy (due to toxicity of nicotine and tobacco products);
* Current alcohol dependence (AUDIT > 15)
* Urine-screened or past-month self-reported use of illicit substances (amphetamine, cocaine, methamphetamine, opioids, benzodiazepines);
* Current psychosis, mania, or suicidal ideation;

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available after the completion of all study activities.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After closing the study IRB protocol and destroying all identifiers. Anticipated 2 years after completion of primary data collection. Data availability will be perpetual. Data dissemination plan is pending.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electronic Cigarette | Smoking As Usual
Started | 12 | 5
Completed Primary Outcome Visit | 11 | 5
Completed | 11 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic Cigarette | Smoking As Usual | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.25 (11.7) | 57.20 (5.26) | 50.88 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 2 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Cigarettes Per Day From Baseline to Week 8 and Week 16
Description: Past week average cigarettes per day assessed using timeline follow-back (TLFB).
Time Frame: Baseline, Week 8, Week 16
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
cigarettes per day
  Baseline | 16.34 (8.68) | 15.39 (6.43)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 9.51 (11.06) | 8.66 (6.83)
  Week 16: number analyzed (Participants) | 11 | 5
  Week 16 | 8.12 (7.06) | 12.30 (10.00)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = .004, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 8.09, 95% CI 2-sided [3.20 to 12.98]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = .060, t-test, 2 sided; Mean Difference (Final Values) = 6.74, 95% CI 2-sided [-0.40 to 13.87] — Paired t-test
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = .766, GEE; Corstr = AR1; test of condition x time interaction; Slope = -.932
Statistical Analysis 4: Comparison: Electronic Cigarette; Repeated measures analysis at Wk 8 and Wk 16 for experimental arm; Test type: Superiority; p = 0.533, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-3.41 to 6.19]
Statistical Analysis 5: Comparison: Smoking As Usual; Repeated measures analysis at Wk 8 and Wk 16 for control arm; Test type: Superiority; p = 0.296, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -3.69, 95% CI 2-sided [-12.21 to 4.84]
Statistical Analysis 6: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.14, GEE; Corstr = AR1; test of condition x time interaction; Slope = -5.075
Statistical Analysis 7: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 16 for experimental arm; Test type: Superiority; p = .002, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 9.48, 95% CI 2-sided [4.24 to 14.71]
Statistical Analysis 8: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = .291, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [-3.91 to 10.01]
Statistical Analysis 9: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = .067, GEE; Corstr = AR1; test of condition x time interaction; Slope = -5.834

2. Primary Outcome: Change in Cigarette Dependence From Baseline to Week 8
Description: Assessed using the Fagerstrom Test for Cigarette Dependence (FTCD). Range: 0-10; higher scores = more dependent.
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
score on a scale
  Baseline | 5.08 (2.68) | 5.60 (2.19)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 4.73 (2.33) | 5.60 (0.89)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = .068, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.07 to 1.71]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 1.00, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0, 95% CI 2-sided [-2.32 to 2.32]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.44, GEE; Corstr = AR1; test of condition x time interaction; Slope = -0.66

3. Primary Outcome: Change in Cigarette Dependence Motives From Baseline to Week 8
Description: Assessed using the Wisconsin Inventory for Smoking Dependence Motives - Brief (Brief-WISDM).
  The value of this outcome variable is the TOTAL SCORE (possible range: 1-7). The TOTAL SCORE is computed as a MEAN of all subscale scores (possible range: 1-7). Each subscale score is the mean of the relevant item scores (possible range: 1-7). Only the TOTAL SCORE is being investigated as an outcome measure.
  HIGHER SCORES = STRONGER dependence motive.
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
score on a scale
  Baseline | 4.79 (0.96) | 5.41 (1.69)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 4.36 (1.56) | 4.18 (2.15)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = .145, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.447, 95% CI 2-sided [-0.184 to 1.078]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 0.280, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-1.50 to 3.95]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.38, GEE; Corstr = AR1; test of condition x time interaction; Slope = .802

4. Primary Outcome: Change in Asthma Symptoms From Baseline to Week 8
Description: Assessed using the Asthma Symptom Utility Index (ASUI). Range: 0-1 continuous; higher scores = fewer or lighter symptoms (0 = worst possible symptoms, 1 = no symptoms).
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
score on a scale
  Baseline | 0.71 (0.18) | 0.65 (0.23)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 0.61 (0.21) | 0.69 (0.23)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = 0.268, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = .086, 95% CI 2-sided [-0.077 to 0.250]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 0.624, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.047, 95% CI 2-sided [-0.291 to 0.198]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.17, GEE; Corstr = AR1; test of condition x time interaction; Slope = -0.15

5. Primary Outcome: Change in Pulmonary Functioning From Baseline to Week 8 (Forced Expiratory Volume [FEV])
Description: Assessed using spirometry and indexed in liters.
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
liters
  Baseline | 2.24 (0.84) | 2.41 (0.53)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 2.32 (0.93) | 2.30 (0.57)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = 0.574, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.077, 95% CI 2-sided [-0.374 to 0.219]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = .077, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [-0.020 to 0.252]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = .149, GEE; Corstr = AR1; test of condition x time interaction; Slope = 0.193

6. Primary Outcome: Change in Pulmonary Functioning From Baseline to Week 8 (Forced Vital Capacity [FVC])
Description: Assessed using spirometry and indexed in liters.
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
liters
  Baseline | 3.02 (1.00) | 3.35 (0.79)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 3.13 (1.16) | 2.98 (0.74)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = 0.376, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.116, 95% CI 2-sided [-0.396 to 0.163]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 0.065, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.036 to 0.78]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = .006, GEE; Corstr = AR1; test of condition x time interaction; Slope = 0.486

7. Primary Outcome: Change in Pulmonary Functioning From Baseline to Week 8 (Forced Expiratory Flow 25%-75% [FEF25-75])
Description: Assessed using spirometry and indexed as liters per section (L/s).
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: liters per second (L/s)
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
liters per second (L/s)
  Baseline | 1.91 (1.00) | 1.82 (0.87)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 1.88 (0.98) | 2.12 (0.64)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = 0.849, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [-0.483 to 0.576]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = .107, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.302, 95% CI 2-sided [-0.706 to 0.102]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.19, GEE; Corstr = AR1; test of condition x time interaction; Slope = -0.34

8. Primary Outcome: Change in Pulmonary Functioning From Baseline to Week 8 (Peak Expiratory Flow [PEF])
Description: Assessed using spirometry and indexed in liters per minute (L/min).
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: liters per minute (L/min)
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
liters per minute (L/min)
  Baseline | 6.50 (2.57) | 6.45 (1.41)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 6.68 (2.91) | 5.69 (1.69)
Statistical Analysis 1: Comparison: Electronic Cigarette; Repeated measures analysis at BL and Wk 8 for experimental arm; Test type: Superiority; p = 0.828, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.085, 95% CI 2-sided [-0.929 to 0.760]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 0.249, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 0.762, 95% CI 2-sided [-0.81 to 2.33]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.17, GEE; Corstr = AR1; test of condition x time interaction; Slope = 0.857

9. Primary Outcome: Change in Fractional Exhaled Nitric Oxide (FENO) From Baseline to Week 8
Description: Level of exhaled FENO assessed with NIOX breath sensor in parts per billion (PPB).
Time Frame: Baseline, Week 8
Population: 1 participant withdrew from the study between baseline and week 8
Measure: Mean (Standard Deviation); unit: parts per billion (PPB)
Arm/Group | Electronic Cigarette | Smoking As Usual
Number analyzed (Participants) | 12 | 5
parts per billion (PPB)
  Baseline | 11.6 (10.2) | 9.80 (8.01)
  Week 8: number analyzed (Participants) | 11 | 5
  Week 8 | 10.9 (8.96) | 7.75 (2.36)
Statistical Analysis 1: Comparison: Electronic Cigarette; Test type: Superiority; p = 0.965, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-9.25 to 8.89]
Statistical Analysis 2: Comparison: Smoking As Usual; Repeated measures analysis at BL and Wk 8 for control arm; Test type: Superiority; p = 0.522, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = 3.25, 95% CI 2-sided [-11.1 to 17.6]
Statistical Analysis 3: Comparison: Electronic Cigarette vs Smoking As Usual; Test type: Superiority; p = 0.781, GEE; Corstr = AR1; test of condition x time interaction; Slope = 1.41

ADVERSE EVENTS:
Time Frame: Entire 8 week experimental and 8 week follow-up period (16 weeks
Description: Adverse changes in medical status were assessed weekly during the experimental period (baseline - wk 8) and again at the final follow-up visit (wk 16)
Arm/Group | Electronic Cigarette | Smoking As Usual
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 1/12 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Cigarette (N=12) | Smoking As Usual (N=5)
Irritation from e-cigarette vapor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Irritation, including coughing, from use of an electronic nicotine delivery system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT05278065/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT05278065/SAP_001.pdf